CLINICAL TRIAL: NCT01614886
Title: A 24-week, Multicenter, Parallel-group, Randomized,Double-blind Study to Evaluate the Tolerability, Safety and Efficacy of 2 Different Titration Methods of Rivastigmine Patch (ENA713D/ONO-2540) in Patients With Mild to Moderate Alzheimer's Disease (MMSE 10-20)
Brief Title: Randomized, Double-blind Study to Evaluate the Tolerability of 2 Different Titration Methods of Rivastigmine Patch in AD Patients (MMSE 10-20)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CENA713D1303
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2015-06

CONDITIONS: Alzheimer's Disease
Keywords: Rivastigmine, Alzheimer's disease, Transdermal patch
MeSH Terms: conditions — Alzheimer Disease | interventions — Rivastigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 step (Experimental)
  Interventions: Drug: Active Comparator
- 3 step (Active Comparator)
  Interventions: Drug: ENA713

INTERVENTIONS:
Drug: Active Comparator — 1-step titration group begin treatment with a rivastigmine patch 9 mg/day for 4 weeks, followed by a dose increase to 18 mg/day.
  Arms: 1 step
Drug: ENA713 — -3-step titration group will begin treatment with a rivastigmine patch 4.5 mg/day for 4 weeks, followed by a further dose increase of 4.5 mg/day at 4-week intervals up to the maintenance dose of 18 mg/day.
  Arms: 3 step

SUMMARY:
To evaluate the tolerability, safety and efficacy of 3-step titration versus 1-step titration of Rivastigmine patch in the Japanese population.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of dementia of the Alzheimer's type according to the DSM-IV criteria
* A clinical diagnosis of probable AD according to NINCDS/ADRDA criteria
* An MMSE score of ≥ 10 and ≤ 20 at baseline

Exclusion Criteria:

* Any medical or neurological conditions other than AD that could explain the patient's dementia
* A current diagnosis of probable or possible vascular dementia
* A score of > 5 on the Modified Hachinski Ischemic Scale (MHIS)
* A current DSM-IV Axis 1 diagnosis that may interfere with the evaluation of the patient's response to study medication.
* Treated with donepezil or galantamine within last 4 weeks before the efficacy assessment at baseline.
* an advanced severe progressive or unstable disease of any type that may interfere with efficacy and safety assessments or put the patient's at special risk
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (43):
- Japan (43):
  - Novartis Investigative Site, Anjo, Aichi-ken
  - Novartis Investigative Site, Ōbu, Aichi-ken
  - Novartis Investigative Site, Seto, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Akita, Akita
  - Novartis Investigative Site, Chiba, Chiba
  - Novartis Investigative Site, Tōon, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Fujioka, Gunma
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Miyoshi, Hiroshima
  - Novartis Investigative Site, Kasama, Ibaraki
  - Novartis Investigative Site, Kamakura, Kanagawa
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kochi, Kochi
  - Novartis Investigative Site, Kōshi, Kumamoto
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Kitamorokata-gun, Miyazaki
  - Novartis Investigative Site, Azumino, Nagano
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Nagaoka, Niigata
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Kanzaki-gun, Saga-ken
  - Novartis Investigative Site, Kasukabe, Saitama
  - Novartis Investigative Site, Kawaguchi, Saitama
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Shizuoka, Shizuoka
  - Novartis Investigative Site, Tokushima, Tokushima
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Koto-ku, Tokyo
  - Novartis Investigative Site, Musashino, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Tachikawa, Tokyo
  - Novartis Investigative Site, Shimonoseki, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Groups:
- Rivastigmine Patch 1 Step: 1-step titration group begins treatment with a rivastigmine patch 9 mg/day for 4 weeks, followed by a dose increase to 18 mg/day
- Rivastigmine Patch 3 Step: 3-step titration group begins treatment with a rivastigmine patch 4.5 mg/day for 4 weeks, followed by a further dose increase of 4.5 mg/day at 4-week intervals up to the maintenance dose of 18 mg/day.
Period: Overall Study
Arm/Group | Rivastigmine Patch 1 Step | Rivastigmine Patch 3 Step
Started | 107 | 109
Safety Population (SAF) | 107 | 108
Full Analysis Set (FAS) | 104 | 105
Completed | 87 | 83
Not Completed | 20 | 26
Not completed — Adverse Event | 15 | 20
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Death | 1 | 0
Not completed — Protocol deviation | 0 | 2

BASELINE CHARACTERISTICS:
Population: Randomized set (RAN) The RAN consisted of all randomized patients. Patients were analyzed according to the treatment group they were assigned to at randomization. A patient was diagnosed of dementia with Lewy Bodies, different from AD, after randomization and was excluded from all analysis (SAF and FAS).
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivastigmine Patch 1 Step | Rivastigmine Patch 3 Step | Total
Number analyzed (Participants) | 107 | 109 | 216
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.5 (6.54) | 77.6 (5.89) | 77.5 (6.21)
Sex/Gender, Customized [Number; unit: Participants] — Baseline characteristics is based on safety analysis set therfore female number is 76.
  Participants
    Female | 69 | 76 | 145
    Male | 38 | 32 | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Adverse Events Leading to Study Drug Discontinuation
Description: The primary variable of this study is the percentage of patients having an AE leading to study drug discontinuation during the 24-week double-blind treatment period.
Time Frame: Up to 24 weeks
Population: Safety population (SAF) This population consisted of all randomized patients who received at least one dose of study medication and had at least one safety assessment after baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivastigmine Patch 1 Step | Rivastigmine Patch 3 Step
Number analyzed (Participants) | 107 | 108
Percentage of participants | 15 | 18.5

2. Secondary Outcome: Change From Baseline in the Alzheimer's Disease Assessment Scale - Japan Cognitive Subscale (ADAS-J Cog)
Description: The Alzheimer's Disease Assessment Scale - Japan cognitive subscale (ADAS-J cog) was used to measure change in cognitive function. The ADAS-J cog score ranges from 0-70, with higher total scores indicating more impairment. A negative change score indicates improvement from baseline.
Time Frame: Baseline, 8,16, and 24 weeks
Population: Full analysis set (FAS): includes all randomized patients who received at least one dose of study drug and had at least one pre- and post-baseline assessment for any of the efficacy variables. n is the number of patients with an assessment at baseline and the corresponding visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rivastigmine Patch 1 Step | Rivastigmine Patch 3 Step
Number analyzed (Participants) | 104 | 105
Units on a scale
  Week 8 (n=99, 100) | -1.3 (3.94) | -0.9 (4.49)
  Week 16 (n=100, 100) | -1.6 (5.01) | -1.2 (5.48)
  Week 24 (n=100, 100) | -1.6 (4.66) | -1.8 (5.58)

3. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE)
Description: The MMSE was used to measure severity of Alzheimer's disease. The test consists of 2 parts: language (time orientation, registration and attention) and performance (recall, response to written/verbal commands, sriting ability and reproduction of complex polygons); the total score can range from 0 to 30, with a higher score indicating better function. A positive change score indicates improvement from baseline.
Time Frame: Baseline and 24 weeks
Population: Full analysis set (FAS): The FAS includes all randomized patients who received at least one dose of study drug and had at least one pre- and post-baseline assessment for any of the efficacy variables. n is the number of patients with an assessment at baseline and the corresponding visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rivastigmine Patch 1 Step | Rivastigmine Patch 3 Step
Number analyzed (Participants) | 94 | 88
Units on a scale | 0.6 (2.91) | 0.5 (3.15)

4. Secondary Outcome: Number of Participants With Improvement in Japanese Clinical Global Impression of Change (J-CGIC). Patients With "Improvement": a Total of 1. Markedly Improved, 2. Improved, and 3. Slightly
Description: The J-CGIC is simple 7 grade investigator's impression scale (1. Markedly improved, 2. Improved, 3. Slightly improved, 4. No change, 5. Slightly aggravated, 6. Aggravated, 7. Markedly aggravated) and a patient is defined to have improvement if J-CGIC tool the values 1, 2, or 3.
Time Frame: 4, 8, 12,16, 20 and 24 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Rivastigmine Patch 1 Step | Rivastigmine Patch 3 Step
Number analyzed (Participants) | 104 | 105
Participants
  Week 4 | 22 | 23
  Week 8 | 35 | 26
  Week 12 | 37 | 33
  Week 16 | 35 | 31
  Week 20 | 32 | 32
  Week 24 | 39 | 38

5. Secondary Outcome: The Percentage of Treatment Retention.
Description: Treatment retention rate at effective dose is defined as the proportion of patients who met all the followings - 1) completed the study, 2) received rivastigmine patch 18 mg/day throughout the last 8 weeks 3) received 18 mg/day for ≥75% of the days during the last 8 weeks
Time Frame: Up to 24 weeks
Population: Safety population (SAF) This population consisted of all randomized patients who received at least one dose of study medication and had at least one safety assessment after baseline. Patients were analyzed according to the treatment group they were assigned to at randomization.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rivastigmine Patch 1 Step | Rivastigmine Patch 3 Step
Number analyzed (Participants) | 107 | 108
Percentage of Participants | 71 | 69.4

ADVERSE EVENTS:
Groups:
- Rivastigmine Patch 1-step: Rivastigmine patch 1-step
- Rivastigmine Patch 3-step: Rivastigmine patch 3-step
Arm/Group | Rivastigmine Patch 1-step | Rivastigmine Patch 3-step
Serious Adverse Events (participants affected / at risk) | 9/107 | 10/108
Other Adverse Events (participants affected / at risk) | 69/107 | 68/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivastigmine Patch 1-step (N=107) | Rivastigmine Patch 3-step (N=108)
Bradycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Dyslalia (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivastigmine Patch 1-step (N=107) | Rivastigmine Patch 3-step (N=108)
Constipation (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 4 | 6
Vomiting (Gastrointestinal disorders) | 5 | 3
Application site dermatitis (General disorders) | 4 | 3
Application site erythema (General disorders) | 17 | 17
Application site pruritus (General disorders) | 24 | 24
Application site rash (General disorders) | 3 | 6
Gastroenteritis (Infections and infestations) | 2 | 3
Influenza (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 9 | 12
Contusion (Injury, poisoning and procedural complications) | 2 | 3
Electrocardiogram QT prolonged (Investigations) | 1 | 3
Weight decreased (Investigations) | 4 | 2
Decreased appetite (Metabolism and nutrition disorders) | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Restlessness (Psychiatric disorders) | 4 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 13 | 12
Eczema (Skin and subcutaneous tissue disorders) | 2 | 3
Hypertension (Vascular disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety